CLINICAL TRIAL: NCT02881008
Title: A Phase 1b/2a Randomized, Open-label Clinical Trial of Daily Myrcludex B Versus Entecavir in Patients With HBeAg Negative Chronic Hepatitis B
Brief Title: Myrcludex B vs Entecavir in Patients With HBeAg Negative Chronic Hepatitis B
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hepatera Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MYR 201 (HBV)
Record Dates: First submitted 2016-08-18; First posted 2016-08-26 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2017-12

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; myrcludex-B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Arm A (Experimental): Myrcludex B 0.5 mg daily for 12 weeks, followed by 12 weeks follow-up period
  Interventions: Drug: Myrcludex B
- Arm B (Experimental): Myrcludex B 1 mg daily for 12 weeks, followed by 12 weeks follow-up period
  Interventions: Drug: Myrcludex B
- Arm C (Experimental): Myrcludex B 2 mg daily for 12 weeks, followed by 12 weeks follow-up period
  Interventions: Drug: Myrcludex B
- Arm D (Active Comparator): Entecavir 0.5 mg daily for 24 weeks
  Interventions: Drug: Entecavir
- Arm E (Experimental): Myrcludex B 5 mg daily for 12 weeks, followed by 12 weeks follow-up period
  Interventions: Drug: Myrcludex B
- Arm F (Experimental): Myrcludex B 10 mg daily for 24 weeks, followed by 12 weeks follow-up period
  Interventions: Drug: Myrcludex B

INTERVENTIONS:
Drug: Entecavir
  Other Names: Baraclude®
  Arms: Arm D
Drug: Myrcludex B
  Other Names: Myrcludex
  Arms: Arm A; Arm B; Arm C; Arm E; Arm F

SUMMARY:
A randomized, open-label multicentre clinical trial of daily Myrcludex B versus entecavir in patients with HBeAg negative chronic hepatitis B.

DETAILED DESCRIPTION:
This is a randomized, open-label multicentre clinical trial of daily Myrcludex B versus entecavir in patients with HBeAg negative chronic hepatitis B. Accounting for screen-outs about 76 patients will be screened and 48 of them will be randomized into 6 treatment groups:

Arm A (8 patients): Myrcludex B 0.5 mg / day / sc / 12 weeks Arm B (8 patients): Myrcludex B 1 mg / day / sc / 12 weeks Arm C (8 patients): Myrcludex B 2 mg / day / sc / 12 weeks Arm D (8 patients): Entecavir 0.5 mg / day / orally / 24 weeks Arm E (8 patients): Myrcludex B 5 mg / day / sc / 12 weeks Arm F (8 patients): Myrcludex B 10 mg / day / sc / 24 weeks

The study consists of screening period up to 28 days (Day -28 -1); baseline visit (Day 0), treatment period up to 12 weeks for groups A-C, E and 24 weeks for groups D, F; follow-up period up to 12 weeks for groups A-C, E, F.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years inclusive at the time of giving of written informed consent for study participation.
2. Chronic hepatitis B defined by the presence of HBsAg for at least 6 months prior to screening period.
3. Liver biopsy performed within one year prior to screening or during screening period.
4. Alanine aminotransferase (ALT) ≥1.5 x ULN and ≤ 6 x ULN. If ALT level during screening period is ≥1 ULN the patient can be included in the study after obtaining the sponsor's approval and if the following conditions are met :

   * evidence of inflammation such as lymphocyte infiltration confirmed by liver biopsy performed within the 6 months prior to the inclusion in the study,
   * and/or the patient has a history of elevated ALT levels of ≥1.5 ULN during the 12 months prior to screening period.
5. HBeAg negative and anti-HBeAg positive.
6. HBV DNA ≥ 104 copies/mL.
7. All women of childbearing potential must have a negative urine pregnancy test prior to enrolment.
8. Women must:

   * Be menopausal for at least 2 years, or
   * Be surgically sterile (total hysterectomy or bilateral ovariectomy or bilateral tubal ligation/clips or otherwise be incapable of pregnancy), or
   * Not be heterosexually active during the study, or
   * Agree to use a highly effective method of birth control (double barrier method or combination of barrier method with hormonal or intrauterine device) during the study and for 3 month after the last dosing of the investigational medicinal product.
9. Men must agree to use a highly effective method of birth control (double barrier methods or combination of barrier method with hormonal or intrauterine device in their women-partner) and not to donate a sperm during the study and for 3 month after the last dosing of the investigational medicinal product.
10. An understanding, ability and willingness to fully comply with study procedures and restrictions.
11. An ability to provide the written informed consent to participate in the study.

Exclusion Criteria:

1. Decompensated liver disease (Child-Pugh-Score >6).
2. Any sign of liver cirrhosis (histological, ultra sound, biochemical).
3. Co-infected with hepatitis C virus (HCV), hepatitis D virus (HDV), or HIV.
4. ALT > 6 ULN.
5. Creatinine clearance < 60 mL/min.
6. Total bilirubin > 2 mg/dL.
7. Pre-treatment with nucleoside-analogues (lamivudine, telbivudine, entecavir) less than 6 months prior to the first dosing of the investigational medicinal products. Pre-treatment with nucleotide-analogues and interferons is allowed.
8. History of hepatocellular carcinoma (HCC) or findings suggestive of possible HCC, such as suspicious foci on imaging studies or elevated serum alpha-fetoprotein (AFP) levels. In patients with such findings, HCC will be ruled-out prior to screening for the present study.
9. One or more additional known primary or secondary causes of liver disease, other than hepatitis B (e.g., alcoholism, autoimmune hepatitis, malignancy with hepatic involvement, hemochromatosis, alpha-1 antitrypsin deficiency, Wilson's Disease, other congenital or metabolic conditions affecting the liver, e.g. congestive heart failure or other severe cardiopulmonary disease). Patients with Gilbert's syndrome and Dubin-Johnson syndrome, two benign disorders associated with low-grade hyperbilirubinemia can be enrolled into the trial.
10. History of clinically evident pancreatitis.
11. History of alcohol or drug abuse within the preceding two years. For the purposes of the present study, alcohol abuse is arbitrarily defined as frequent consumption of alcoholic beverages with an average daily intake of more than 40 g of ethanol.
12. Participation in another study with an investigational drug within less than one month prior to this study or simultaneously to this study.
13. Patients who are unable or unwilling to follow the protocol requirements.
14. Patients with a history of seizures, central nervous system disorders or psychiatric disability thought to be clinically significant in the opinion of the investigator.
15. Patients with limited mental capacity to the extent that she/he cannot provide informed consent or information regarding adverse events of the study drug.
16. Clinically significant renal, respiratory or cardiovascular disease.
17. Pregnancy and lactation.
18. Patients who have previously participated in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-11-14 (Actual); Primary Completion 2014-10-04 (Actual); Study Completion 2014-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Bogomolov, PhD, Principal Investigator — LLC "Clinical Hospital of Tsentrosoyuz"
Locations (9):
- Russia (9):
  - SBEI of Higher Professional Education "South Ural State Medical university" of the MoH of the RF, Chelyabinsk
  - 1-st MMU n.a. I.M. Sechenov based in Moscow State-Owned Health Care Institution "Infectious Clinical Hospital № 2 of Moscow Healthcare Department", Moscow
  - FSBI of Higher Education "People's Friendship University", Moscow
  - FSBHI "Central Clinical Hospital RAS", Moscow
  - LLC "Clinical Hospital of Tsentrosoyuz", Moscow
  - SPb SBHI "The Center for Prevention and Control of AIDS and Infectious Diseases", Saint Petersburg
  - SPb SIH "Clinical Centre of Infectious Diseases Named After S.P. Botkin", Saint Petersburg
  - Medical Company "Hepatolog" LLC, Samara
  - SBIH "Stavropol Regional Clinical Hospital", Stavropol

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lavanchy D. Hepatitis B virus epidemiology, disease burden, treatment, and current and emerging prevention and control measures. J Viral Hepat. 2004 Mar;11(2):97-107. doi: 10.1046/j.1365-2893.2003.00487.x. PMID 14996343
- [Background] Yan H, Zhong G, Xu G, He W, Jing Z, Gao Z, Huang Y, Qi Y, Peng B, Wang H, Fu L, Song M, Chen P, Gao W, Ren B, Sun Y, Cai T, Feng X, Sui J, Li W. Sodium taurocholate cotransporting polypeptide is a functional receptor for human hepatitis B and D virus. Elife. 2012 Nov 13;1:e00049. doi: 10.7554/eLife.00049. PMID 23150796
- [Background] Trauner M, Boyer JL. Bile salt transporters: molecular characterization, function, and regulation. Physiol Rev. 2003 Apr;83(2):633-71. doi: 10.1152/physrev.00027.2002. PMID 12663868
- [Background] Lok AS, McMahon BJ. Chronic hepatitis B: update 2009. Hepatology. 2009 Sep;50(3):661-2. doi: 10.1002/hep.23190. No abstract available. PMID 19714720
- [Background] Nowak MA, Bonhoeffer S, Hill AM, Boehme R, Thomas HC, McDade H. Viral dynamics in hepatitis B virus infection. Proc Natl Acad Sci U S A. 1996 Apr 30;93(9):4398-402. doi: 10.1073/pnas.93.9.4398. PMID 8633078
- [Background] Yan H, Zhong G, Xu G, He W, Jing Z, Gao Z, Huang Y, Qi Y, Peng B, Wang H, Fu L, Song M, Chen P, Gao W, Ren B, Sun Y, Cai T, Feng X, Sui J, Li W. Sodium taurocholate cotransporting polypeptide is a functional receptor for human hepatitis B and D virus. Elife. 2012 Nov 13;3. doi: 10.7554/eLife.00049. PMID 25409679

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F
Started | 8 | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population - all randomized patients who were administered at least one dose of the study drugs.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (8.5) | 32.9 (10.6) | 42.4 (11.1) | 40.2 (13.0) | 36.4 (9.5) | 34.5 (6.7) | 37.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 4 | 3 | 2 | 16
  Male | 5 | 7 | 5 | 4 | 5 | 6 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 7 | 8 | 8 | 8 | 7 | 8 | 46
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russia | 8 | 8 | 8 | 8 | 8 | 8 | 48

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With HBsAg Response at 12 Week of Therapy
Description: HBsAg response is defined as serum HBsAg decline of at least 0.5 logs IU/ml (or HBsAg negativation) at week 12 compared to baseline.
Time Frame: 12 week
Population: For the efficacy assessments the main analysis set was Full analysis set (FAS): All patients of the Safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
Participants | 0 | 0 | 1 | 0 | 0 | 0

2. Secondary Outcome: Proportion of Patients With HBsAg Response at 24 Week of Therapy
Description: HBsAg response is defined as serum HBsAg decline of at least 0.5 logs IU/ml (or HBsAg negativation) at week 24 compared to baseline.
Time Frame: 24 weeks
Population: This variable was assessed in the patients administered 24-week treatment: patients of Arm F who received Myrcludex B 10 mg and patients of Arm D who received Entecavir 0.5 mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm D | Arm F
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

3. Secondary Outcome: Proportion of Patients With HBV DNA Response at Week 12 of Therapy
Description: HBV DNA response is defined as persistent reduction of HBV DNA by >1 log IU/ml or negativation at week 12 compared to baseline.
Time Frame: 12 weeks
Population: For the efficacy assessments the main analysis set was Full analysis set (FAS): All patients of the Safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
Participants | 2 | 0 | 2 | 8 | 1 | 6

4. Secondary Outcome: Proportion of Patients With Biochemical Response at 12 Weeks of Therapy
Description: Biochemical response is defined as normalization of ALT level at week 12 compared to baseline.
Time Frame: 12 weeks
Population: Only patients with abnormal ALT levels at baseline were included in data analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F
Number analyzed (Participants) | 7 | 7 | 8 | 7 | 4 | 6
Participants | 3 | 4 | 4 | 4 | 2 | 4

5. Secondary Outcome: Proportion of Patients With cccDNA Response at 24 Week of Therapy
Description: Virological cccDNA response is defined as reduction of intrahepatic cccDNA by 0.5 logs in comparison to baseline at week 24.
Time Frame: 24 weeks
Population: Virological cccDNA response was to be estimated only for patients of group F administered 24-week therapy with Myrcludex B in the dose of 10 mg and to whom liver biopsy during screening period and at week 24 was performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm F
Number analyzed (Participants) | 5
Participants | 0

6. Secondary Outcome: Proportion of Patients With HBV DNA Response at Week 24 of Therapy
Description: HBV DNA response is defined as persistent reduction of HBV DNA by >1 log IU/ml or negativation at week 24 compared to baseline.
Time Frame: 24 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm D | Arm F
Number analyzed (Participants) | 8 | 8
Participants | 7 | 6

7. Secondary Outcome: Proportion of Patients With Biochemical Response at 24 Weeks of Therapy
Description: Biochemical response is defined as normalization of ALT level at week 24 compared to baseline.
Time Frame: 24 weeks
Population: This variable was assessed in the patients administered 24-week treatment: patients of Arm F who received Myrcludex B 10 mg and patients of Arm D who received Entecavir 0.5 mg. Only patients with abnormal ALT levels at baseline were included in data analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm D | Arm F
Number analyzed (Participants) | 7 | 6
Participants | 5 | 3

ADVERSE EVENTS:
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/8 | 1/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 6/8 | 5/8 | 2/8 | 4/8 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=8) | Arm B (N=8) | Arm C (N=8) | Arm D (N=8) | Arm E (N=8) | Arm F (N=8)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=8) | Arm B (N=8) | Arm C (N=8) | Arm D (N=8) | Arm E (N=8) | Arm F (N=8)
Eosinophilia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site dermatitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reticulocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Xeroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other